CLINICAL TRIAL: NCT04213742
Title: Study on the Application of Gratitude Intervention in Patients With Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KY20192028-F-2
Record Dates: First submitted 2019-12-24; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Patients ； Spinal Cord Injury

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gratitude diary (Active Comparator)
  Interventions: Other: Thanksgiving diary intervention
- No intervention (No Intervention)
- Gratitude visit (Active Comparator)
  Interventions: Other: Thanksgiving diary intervention

INTERVENTIONS:
Other: Thanksgiving diary intervention — Record gratitude.
  Arms: Gratitude diary; Gratitude visit

SUMMARY:
To analyze the present situation and influencing factors of gratitude level and quality of life of patients with spinal cord injury, and to explore the methods of Thanksgiving intervention for patients with spinal cord injury so as to provide scientific basis for improving the quality of life of patients with spinal cord injury.

Investigation and research design and experimental research design

DETAILED DESCRIPTION:
Effectiveness evaluation indicators: (1) main efficacy indicators: gratitude level scale (C-GQ-6) score, quality of life scale (WHOQOL-BREF) score; (2) secondary efficacy index: positive psychological capital scale (PPQ) score; trait coping style (TCSQ) score, perceived social support scale (PSSS) score.

Inclusion criteria: accorded with the 6th edition of neurological classification of spinal cord injury issued by the American Spinal Cord injury Society, and confirmed by CT or MRI imaging; sequelae such as limb motor dysfunction caused by spinal cord injury; age ≥ 18 years old; returned to the community after discharge from hospital for at least 2 weeks; good language communication skills, volunteered to participate in this study; Exclusion criteria: spinal cord injury caused by non-trauma (such as bone tumor, spinal cord angiopathy, medical operation, etc.); patients with brain organic diseases; those who were diagnosed with mental disorders; unwilling to participate in this researcher;

ELIGIBILITY:
Inclusion Criteria:

* Conformed to the 6th edition of neurological classification of spinal cord injury issued by the American Spinal Cord injury Society, and confirmed by CT or MRI imaging; sequelae such as different degrees of limb motor dysfunction caused by spinal cord injury; age ≥ 18 years old; returned to the community after discharge from the hospital for at least 2 weeks; good language communication skills, volunteered to participate in this study;

Exclusion Criteria:

* Non-traumatic spinal cord injury (such as bone tumor, spinal cord angiopathy, medical operation, etc.); patients with brain organic diseases; those with definite diagnosis of mental disorders; unwilling to participate in this researcher;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Gratitude scale (GQ-6) ； | 5 minutes
  The scale consists of 6 items and is graded at Likert7 level.
Quality of life scale (WHOQOL-BREF) ； | 5 minutes
  The scale consists of 26 items and 4 dimensions, namely, self-efficacy, resilience, hope and optimism, which are used to measure the level of individual psychological capital, using Likert7 score.
Positive psychological capital scale (PPQ) | 5 minutes
  The scale consists of 26 items and 4 dimensions, namely, self-efficacy, resilience, hope and optimism, which are used to measure the level of individual psychological capital, using Likert7 score.

CONTACTS AND LOCATIONS:
Locations (1):
- 第四军医大学, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided